CLINICAL TRIAL: NCT04661501
Title: The BREAST Trial: A Randomized, Non-inferiority, Study Comparing the Complication Profile of Four Commercially Available Acellular Dermal Matrixes Used in Alloplastic Breast Reconstruction
Brief Title: BREAST ADM Trial for Alloplastic Breast Reconstruction
Acronym: Breast_ADM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Nancy Van Laeken, Clinical Professor, Division of Plastic Surgery, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H18-02052
Record Dates: First submitted 2020-10-23; First posted 2020-12-10 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Breast Reconstruction

STUDY DESIGN:
Who Masked: Participant
Masking Description: Treatment information will be non-blinded to the surgical staff who will then proceed to order the appropriate ADM product to be available at the time of the study participants scheduled breast reconstruction. Additionally, randomization will occur independently for each surgeon prevent bias from arising as a result of the surgeon performing the reconstruction.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AlloDerm group (Active Comparator): Device for immediate implant based breast reconstruction.
  Interventions: Device: AlloDerm
- AlloMax group (Active Comparator): Device for immediate implant based breast reconstruction.
  Interventions: Device: AlloMax
- DermACELL group (Active Comparator): Device for immediate implant based breast reconstruction.
  Interventions: Device: DermACELL
- Flex HD group (Active Comparator): Device for immediate implant based breast reconstruction.
  Interventions: Device: Flex HD

INTERVENTIONS:
Device: AlloDerm — Acellular Dermal Matrices (ADMs) are breast reconstruction material. They are donated cadaveric dermis that is aseptically processed or sterilized in order to remove cellular and immunogenic components to prevent host reactions.
  Arms: AlloDerm group
Device: AlloMax — Acellular Dermal Matrices (ADMs) are breast reconstruction material. They are donated cadaveric dermis that is aseptically processed or sterilized in order to remove cellular and immunogenic components to prevent host reactions.
  Arms: AlloMax group
Device: DermACELL — Acellular Dermal Matrices (ADMs) are breast reconstruction material. They are donated cadaveric dermis that is aseptically processed or sterilized in order to remove cellular and immunogenic components to prevent host reactions.
  Arms: DermACELL group
Device: Flex HD — Acellular Dermal Matrices (ADMs) are breast reconstruction material. They are donated cadaveric dermis that is aseptically processed or sterilized in order to remove cellular and immunogenic components to prevent host reactions.
  Arms: Flex HD group

SUMMARY:
This study is a randomized single blinded prospective clinical trial comparing the surgical outcomes of four different acellular dermal matrixes (ADMs) after primary breast reconstruction. ADMs are used in conjunction with tissue expanders or breast implants to reinforce the recreated breast pocket. Currently, 4 different ADMS are commercially available: AlloDerm, DermaCell, Allomax and Flex HD. It is unclear which ADM is clinically superior. The objective of the study is to compare the complications and post-op care of 4 different ADMs within a 2 year follow up to elucidate their surgical outcomes.

DETAILED DESCRIPTION:
This study is a randomized control trial and will include all patients who are agreeable and deemed appropriate for alloplastic breast reconstruction involving the use of an ADM with two stage tissue expander (TE) reconstruction. The ADMs used will be determined by random assignment to one of four available products being utilized within the study: AlloDerm, AlloMax, DermACELL and FlexHD. Each ADM product will comprise of an individual treatment arm. Participants undergoing bilateral reconstruction will have the same ADM used in each side. The four treatment arms will be compared to assess their impact on our primary outcome: proportion of clinically significant post-operative seroma requiring intervention. Analysis will be performed per surgeon to prevent post-operative outcomes from being confounded by the principle operator. The trial will initially be conducted as an internal pilot study. The study will initially target a study population of 40 patients for recruitment as a means to assess the feasibility of the study. In doing this, the pilot study will be able to establish the necessary protocol and administrative infrastructure that is needed to complete the trial in its entirety. This create a sample population for initial outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All woman aged 21 years or older but less that 65 undergoing unilateral or bilateral mastectomy with alloplastic breast reconstruction using ADM.
* Breast reconstruction must be done by means of a two staged process using tissue expanders and ADM based reconstruction followed by implant tissue expander to implant exchange.

Exclusion Criteria:

* Patients undergoing autologous reconstruction either at the time of mastectomy or in a delayed fashion.
* Patients with a history of previous breast reconstruction procedures.
* Patients with prior radiation treatment to the breast or with prior mantle radiation
* Any patient with a contraindication to breast reconstruction
* Patients undergoing an axillary node dissection with clearance
* Patients with an allergy to Polysporin or any of its ingredients.
* Patients with contraindications to any of the acellular dermal matrices:

  • DermACELL: Allergy to Gentamicin, Vancomycin[12]
* The surgeon performing the breast reconstruction may also deem a patient ineligible if intraoperatively, there is evidence of significant mastectomy flap ischemia prior to the initiation of the breast reconstruction procedure.

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Seroma incidence | Within 6 months of stage I or stage II surgery
  Incidence of seroma formation requiring intervention including aspiration in-office or ultrasound-guided drainage

SECONDARY OUTCOMES:
Mean drain duration (Days) | Within 1 month of stage I or stage II surgery
  Postoperative duration of drain placements
Mean drain output (ml) | Within 1 month of stage I or stage II surgery
  Total volume of drain output until drain removal
Mean seroma volume (ml) | Within 6 months of stage I or stage II surgery
  Total volume of seroma fluid aspirated until resolution of seroma
Mean aspirations per seroma | Within 6 months of stage I or stage II surgery
  Number of aspirations required for seroma resolution
Hematoma incidence | Within 1 month of stage I or stage II surgery
  Incidence of hematoma requiring evacuation or aspiration
Surgical site infection incidence | Within 6 months of stage I or stage II surgery
  Incidence of surgical site infection requiring antibiotics or operative management
Number of Participants with Implant loss | Within 2 year of stage II surgery
  Loss of Implant for any reason (wound dehiscence, exposure, periprosthetic infection)
Number of Participants with Red breast syndrome | Within 1 month of stage I surgery
  Noninfectious erythema localized to the area of ADM reconstruction
Number of Participants with Unplanned surgical care | Within 2 year of stage I or stage II surgery
  Unexpected return to the operating room that was not planned at the initial visit for any reason
Number of Participants with Mastectomy flap necrosis | Within 1 month of stage I surgery
  Mastectomy flap necrosis and associated management: expectant, office debridement, or return to the operating room
Capsular contracture incidence | Within 1 year of stage II surgery
  Incidence of capsular contracture (as identified by the plastic surgeon, grouped by Baker's classification of severity)
ADM integration assessment | Within 1 month of stage II procedure
  Clinical assessment of ADM integration into the breast pocket at the time of the second stage procedure.
Post-operative aesthetic assessment (patient and surgeon) | Within 2 years of stage II surgery
  Subjective assessment of cosmetic outcome by the patient and blinded assessors using post-operative aesthetic breast survey assessment
Pre and post-operative satisfaction assessed using BREAST-Q | Within 2 years of stage II surgery
  Evaluation of the satisfaction and quality of life of patients undergoing breast surgery using the BREAST-Q. Breast-Q is based on Breast Cancer Core Scale ranging from 0 to 100. Higher score means better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nancy Van Laeken, Principal Investigator — University of British Columbia
Locations (4):
- Canada (4):
  - Mount Saint Joseph's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - UBC Hospital, Vancouver, British Columbia
  - Saint Paul's Hospital, Vancouver, British Columbia

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/01/NCT04661501/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/01/NCT04661501/ICF_001.pdf